CLINICAL TRIAL: NCT06045767
Title: T-Cell Repertoire Sequencing: Assessing Pembrolizumab Efficacy in Advanced Non-small Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ari Raphael (Other)
Collaborators: Bar-Ilan University, Israel (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Ari Raphael, Head Oncology Day-care unit, Tel Aviv Medical Center
Organization: Tel Aviv Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0222-24 TLV
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Non-small Cell Lung Cancer Metastatic
Keywords: T-cell repertoire; ctDNA
MeSH Terms: interventions — pembrolizumab; Injections; Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pembrolizumab + Carboplatin+ Pemetrexed (Experimental)
  Interventions: Drug: Pembrolizumab 50 MG Injection [Keytruda]

INTERVENTIONS:
Drug: Pembrolizumab 50 MG Injection [Keytruda] — Chemo-immunotherapy combination
  Other Names: Carboplatin; Pemetrexed

SUMMARY:
This is a single site, non-randomized trial for the assessment of intravenous (IV) pembrolizumab (also known as MK-3475) combined with pemetrexed/platinum-based chemotherapy in subjects with advanced or metastatic non-squamous non-small lung cancer (NSCLC) who have not previously received systemic therapy for advanced disease and in whom directed therapy is not indicated. Approximately 30 subjects will be enrolled in this trial to examine the clonality and diversity dynamics matched with disease response evaluated by RECIST 1.1.

DETAILED DESCRIPTION:
Subjects will receive pembrolizumab 200 mg combined with pemetrexed and platinum (investigator's choice of cisplatin or carboplatin), as indicated below:

Pembrolizumab 200 mg + pemetrexed 500 mg/m2 (with vitamin supplementation) + cisplatin 75 mg/m2 OR carboplatin AUC 5, all on Day 1 every 3 weeks (Q3W) for 4 cycles followed by pembrolizumab 200 mg + pemetrexed 500 mg/m2 Q3W until progression.

Treatment with pembrolizumab and pemetrexed will continue until 35 trial treatments have been administered, documented disease progression or unacceptable adverse event(s).

Patients will be stratified according to clinical and histopathological parameters: 1. PD-L1 status (PD-L1 >/= 1 or <1) 2. Age < 65 vs => 65 3. Smoking history yes vs no 4. Platinum chemotherapy: cisplatin vs. carboplatin 5. Immune-related adverse events (irAEs).

TCR repertoire clonality and diversity will serve as an assessment measure for treatment response, along with PET/CT-scans, tumor exomal profile and ctDNA dynamics.

ELIGIBILITY:
Inclusion Criteria:

* Participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
* Have measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Archival tumor tissue sample or newly obtained [core, incisional or excisional] biopsy of a tumor lesion not previously irradiated has been provided.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Adequate organ function.

Exclusion Criteria:

* Pregnancy or breastfeeding
* Aberration in a known targetable molecular driver.
* Received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor.
* Received prior systemic anti-cancer therapy for metastatic disease.
* Received prior radiotherapy within 2 weeks of start of study intervention.
* Major surgery within 14 days.
* Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy.
* Known additional malignancy that is progressing or has required active treatment within the past 3 years.
* Known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated or asymptomatic brain metastases may participate provided they are radiologically stable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) per RECIST 1.1 - correlated to TCR repertoire data, such as clonality/diversity. | 5 years
  ORR defined as the percentage of participants who achieve a confirmed complete response (CR) or partial response (PR) per RECIST 1.1 as assessed by the investigator.
  By integrating serial TCR repertoire sequencing (Rep-seq) of NSCLC patients treated with pembrolizumab and platinum-based chemotherapy regimens we aim to capture the temporal clonality and diversity dynamics with the disease response.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) correlated with circulating tumor DNA (ctDNA), by measurement of variant allele frequency (VAF). | 5 years
  To capture the VAF in ctDNA, and correlate it with response to therapy evaluated by ORR per RECIST 1.1. We will capture its dynamics throughout blood samples collected longitudinally (pre-and during treatment).

CONTACTS AND LOCATIONS:
Overall Officials: Ari Raphael, M.D, Principal Investigator — Tel-Aviv University school of medicine